CLINICAL TRIAL: NCT04418323
Title: Video-assisted Anal Fistula Treatment (VAAFT) Versus Fistula-tract Laser Closure (Filac) Versus Conventional Seton in the Management of Anal Fistula
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R.19.03.453 - 2019/03/11
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-05

CONDITIONS: Video Assisted Anal Fistula Treatment

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Video-assisted anal fistula treatment (VAAFT (Active Comparator): Video-assisted anal fistula treatment (VAAFT) in the Management of anal fistula
  Interventions: Procedure: Video-assisted anal fistula treatment (VAAFT) versus Fistula-tract Laser Closure (filac) versus Conventional seton in the Management of anal fistula
- Fistula-tract Laser Closure (filac) (Active Comparator): Fistula-tract Laser Closure (filac)in the Management of anal fistula
  Interventions: Procedure: Video-assisted anal fistula treatment (VAAFT) versus Fistula-tract Laser Closure (filac) versus Conventional seton in the Management of anal fistula
- Conventional seton (Active Comparator): Conventional seton in the Management of anal fistula
  Interventions: Procedure: Video-assisted anal fistula treatment (VAAFT) versus Fistula-tract Laser Closure (filac) versus Conventional seton in the Management of anal fistula

INTERVENTIONS:
Procedure: Video-assisted anal fistula treatment (VAAFT) versus Fistula-tract Laser Closure (filac) versus Conventional seton in the Management of anal fistula — Video-assisted anal fistula treatment (VAAFT) versus Fistula-tract Laser Closure (filac) versus Conventional seton in the Management of anal fistula

SUMMARY:
Anal fistula is a chronic inflammatory tract connecting an internal opening in the anal canal with one or more than one external openings in the perianal skin Aim of the work This prospective randomized control trial, we will compare video-assisted anal fistula treatment (Vaaft) and Fistula Laser closure (Filac) and conventional Seton as regards, recurrence rate as a primary outcome. Secondary outcome includes; operative and post-operative data, hospital stay, pain score, healing time, return to work and continence

ELIGIBILITY:
Inclusion Criteria:

* Patients of both genders aging between 18-65 years with cryptoglandular anal fistula will be included.

Exclusion Criteria:

* We will exclude patients with associated anorectal pathology such as anal fissure, hemorrhoids, rectal prolapse, neoplasm, solitary rectal ulcer, inflammatory bowel diseases, and patients on long acting corticosteroids or immunosuppressive drugs will be also excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-06-16 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-02 (Estimated)

PRIMARY OUTCOMES:
recurrence of anal fistula | one year
  recurrence of anal fistula symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt